CLINICAL TRIAL: NCT02171507
Title: Relative Bioavailability of Dabigatran and Diclofenac After 150 mg b.i.d. Dabigatran Etexilate and Diclofenac at 50 mg Single Dose Alone or Following Concomitant Multiple Oral Administrations in Healthy Male and Female Volunteers (an Open Label, Randomised, Multiple- Dose, Three-way Crossover Study)
Brief Title: Relative Bioavailability of Dabigatran and Diclofenac After Dabigatran Etexilate and Diclofenac Single Dose Alone or Following Concomitant Multiple Oral Administrations in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.7
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Diclofenac

ARMS (3):
- Dabigatran etexilate (Active Comparator)
  Interventions: Drug: Dabigatran etexilate
- Diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac
- Dabigatran etexilate + diclofenac (Experimental)
  Interventions: Drug: Dabigatran etexilate; Drug: Diclofenac

INTERVENTIONS:
Drug: Dabigatran etexilate
  Arms: Dabigatran etexilate; Dabigatran etexilate + diclofenac
Drug: Diclofenac
  Arms: Dabigatran etexilate + diclofenac; Diclofenac

SUMMARY:
To investigate the relative bioavailability of dabigatran with and without concomitant administration of diclofenac and the relative bioavailability of diclofenac with and without concomitant administration of dabigatran etexilate

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, clinical laboratory tests
2. Age ≥18 and ≤55 years
3. Body mass index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion criteria:

1. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder including history of gastrointestinal erosions and ulcer or acute blood coagulation defect
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the objectives of the trial as judged by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance
16. Subjects with abnormal thrombocyte counts and any relevant deviation in the assessment of platelet function (PFA test) must be excluded
17. Inability to comply with dietary regimen of study centre
18. Females of child bearing potential who are pregnant, breast feeding or who are either not surgically sterile or are sexually active and not using an acceptable form of contraception as either the oral contraceptives since at least two months and the double barrier method, i.e. intrauterine device with spermicide and condom for the male partner
19. Male subjects must agree to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the post study medical examination. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)
20. Planned surgeries within four weeks following the end-of study examination
21. Intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, cumarin etc.
22. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
23. Vulnerable subjects (e.g. persons kept in detention).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss on Day 4 (area under the concentration-time curve of dabigatran in plasma at steady state over one dosing interval) | from pre-dose up to 72 hours post-dose
Cmax,ss (maximum concentration of dabigatran in plasma at steady state) | from pre-dose up to 72 hours post-dose
Cmax (maximal concentration of diclofenac in plasma) | from pre-dose up to 72 hours post-dose
AUC0-infinity (area under the concentration-time curve of diclofenac in plasma extrapolated to infinity) | from pre-dose up to 72 hours post-dose
aPTT (activated partial thromboplastin time) and ECT (Ecarin clotting time) with and without diclofenac | from pre-dose up to 72 hours post-dose
AUERτ,ss (area under the effect ratio-time curve of dabigatran in plasma at steady state over a uniform dosing interval τ) | from pre-dose up to 72 hours post-dose
ERmax,ss (maximal effect ratio of dabigatran in plasma at steady state) | from pre-dose up to 72 hours post-dose

SECONDARY OUTCOMES:
AUC0-tz,ss (area under the concentration-time curve of dabigatran in plasma from the time point 0 after the last dose at steady state to the last quantifiable dabigatran plasma concentration within the uniform dosing interval τ) | from pre-dose up to 72 hours post-dose
tz,ss (time of last measurable concentration of dabigatran in plasma within the dosing interval τ at steady state) | from pre-dose up to 72 hours post-dose
tmax,ss (time from last dosing to the maximum concentration of dabigatran in plasma at steady state on Day 4) | from pre-dose up to 72 hours post-dose
CL/Fss (apparent clearance of dabigatran in the plasma at steady state after extravascular multiple dose administration) | from pre-dose up to 72 hours post-dose
CLR,ss (renal clearance of dabigatran at steady state determined over the dosing interval τ) | from pre-dose up to 72 hours post-dose
C min,ss (minimum measured concentration of dabigatran in plasma at steady state over a uniform dosing interval τ) | from pre-dose up to 72 hours post-dose
tmin,ss (time from last dosing to the minimum concentration of dabigatran in plasma at steady state over a uniform dosing interval τ) | from pre-dose up to 72 hours post-dose
Cpre,ss (pre-dose concentration of dabigatran in plasma at steady state immediately before administration of the next dose) | from pre-dose up to 72 hours post-dose
MRTp.o.,ss (mean residence time of dabigatran in the body at steady state after oral administration) | from pre-dose up to 72 hours post-dose
Vz/Fss (apparent volume of distribution during the terminal phase λz at steady state following an extravascular administration) | from pre-dose up to 72 hours post-dose
Aeτ,ss (amount of dabigatran that is eliminated in urine at steady state over a uniform dosing interval τ) | 0 to 12 h and 12 to 24 h after administration on day 4
feτ,ss (fraction of parent drug eliminated in urine at steady state over a uniform dosing interval τ) | 0 to 12 h and 12 to 24 h after administration on day 4
AUC0-tz (area under the concentration-time curve of diclofenac and 4´- hydroxydiclofenac in plasma over the time interval 0 to the last quantifiable analyte plasma concentration after single dose administration) | from pre-dose up to 72 hours post-dose
tz (time of last measurable concentration of diclofenac and 4´- hydroxydiclofenac in plasma following a single dose) | from pre-dose up to 72 hours post-dose
%AUCtz-infinity (percentage of the AUC0-infinity that is obtained by extrapolation) for diclofenac and 4´- hydroxydiclofenac | from pre-dose up to 72 hours post-dose
tmax (time from dosing to the maximum concentration of diclofenac and 4´- hydroxydiclofenac in plasma following a single dose) | from pre-dose up to 72 hours post-dose
λz (terminal rate constant in plasma after a single dose) for diclofenac and 4´- hydroxydiclofenac | from pre-dose up to 72 hours post-dose
t1/2 (terminal half-life of diclofenac and 4´- hydroxydiclofenac in plasma after a single dose) | from pre-dose up to 72 hours post-dose
MRTp.o. (mean residence time of diclofenac and 4´- hydroxydiclofenac in the body after single dose oral administration) | from pre-dose up to 72 hours post-dose
CL/F (apparent clearance of diclofenac and 4´- hydroxydiclofenac in the plasma after extravascular single dose administration) | from pre-dose up to 72 hours post-dose
Vz/F (apparent volume of distribution during the terminal phase λz following extravascular dose) for diclofenac and 4´- hydroxydiclofenac | from pre-dose up to 72 hours post-dose